CLINICAL TRIAL: NCT07290205
Title: Neuroimaging of Sedation With Remimazolam
Brief Title: Remimazolam NeuroImaging
Acronym: REMAZ
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Keith M Vogt (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor-Investigator, Keith M Vogt, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY25110017; R35GM146822 (NIH)
Record Dates: First submitted 2025-12-12; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Anesthesia; Pain; Remimazolam
Keywords: Remimazolam; functional MRI; electric nerve stimulation; sedation; functional connectivity; memory; pain
MeSH Terms: conditions — Pain | interventions — remimazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Remimazolam+Pain (Experimental): Single-arm study. All subjects receive remimazolam and painful electric nerve stimulation, while being imaged with MRI, as described in the interventions.
  Interventions: Drug: Remimazolam; Device: Peripheral Nerve Stimulation

INTERVENTIONS:
Drug: Remimazolam — Subjects in this group will receive an intravenous infusion of this drug, during a portion of the study.
Device: Peripheral Nerve Stimulation — Experimental acute pain stimulus will be delivered using a nerve stimulator. These painful shocks will be paired with a fixed number of the experimental cues, in a pattern that appears random to participants.

SUMMARY:
This is a single-arm functional MRI study that will determine the effects of remimazolam on cognition and brain activity and connectivity at rest, during noxious stimulation, and during a memory encoding task

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-59 years of age, who:
* have none of the specific exclusion criteria
* have a valid email address and valid phone number throughout the study
* free from any non-MRI compatible implants

Exclusion Criteria:

* are pregnant or attempting to conceive
* body mass index (BMI) > 35
* significant memory impairment or hearing loss
* sleep apnea
* chronic pain or frequently taking pain medication (including tramadol)
* chronic medical conditions requiring treatment (hypertension, diabetes, high cholesterol)
* neurologic disease, including seizures and tremor
* psychiatric diagnoses, including anxiety, depression, panic, or PTSD
* a history of any of these medical conditions: abnormal heartbeats (cardiac conduction abnormality or arrhythmia), liver or kidney disease, or significant lung disease
* severe claustrophobia or MRI intolerance
* have metal implants or non-removable metal piercings
* having a history of adverse reaction to midazolam (Versed), lorazepam (Ativan) or another benzodiazepine class medication
* are allergic to dextran
* daily alcohol or heavy alcohol use; history of alcohol abuse
* current daily smoker
* regular or recent marijuana use (including prescribed/medical marijuana)
* illicit drug use, i.e., street drugs
* regularly taking: antiepileptics, antidepressants, anti-psychotics, antihistamines, anti-anxiety medication, stimulants, or sleep-aids

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-02 (Estimated)

PRIMARY OUTCOMES:
Explicit memory performance | Day/Visit 2: 12-36 hours after day 1 session
  Recognition memory testing, using the Remember-Know procedure, in which subjects indicate whether they recognize previously experienced experimental items among novel items (not previously in the experiment). This allows calculation of interdependent measures of recollection & familiarity using the signal detection statistic, d'. d' is calculated as the cumulative Gaussian distribution of false positive responses subtracted from the cumulative Gaussian distribution of correctly identified previously-experienced items. d' is on a (theoretically infinite) scale of standard deviation units, with negative values representing performance worse than chance guessing and positive values representing stand deviations of performance above chance. Cross-condition comparisons will be the main effect of interest, comparing no drug to remimazolam.
subjective pain ratings | Day/Visit 1: immediately after no-drug condition MRI scan and immediately after remimazolam condition MRI scan
  Numerical ratings of pain intensity and unpleasantness will be obtained after each experimental period involving repeated noxious stimulation. Values will be on a 0-10 scale, with 0 representing none and 10 representing the worst possible rating.

SECONDARY OUTCOMES:
functional magnetic resonance imaging activation of memory encoding task | Day/Visit 1: during no-drug condition MRI scan and during remimazolam MRI scan
  Event-related blood-oxygen level dependent (BOLD) Magnetic Resonance Imaging (MRI) responses will be determined for each experimental item presented, revealing localized changes in blood flow, which correlate to increased neuronal activity. These will be averaged across the multiple repetitions of memory-encoding experimental events, creating an anatomical map of Z-scores. Cross-condition comparisons will be the main effect of interest, comparing no drug to remimazolam.
functional magnetic resonance imaging activation of the response to noxious stimulation | Day/Visit 1: during no-drug condition MRI scan and during remimazolam MRI scan
  Event-related blood-oxygen level dependent (BOLD) Magnetic Resonance Imaging (MRI) responses will be determined for each experimental item presented, revealing localized changes in blood flow, which correlate to increased neuronal activity. These will be averaged across the multiple repetitions of noxious stimulation events, creating an anatomical map of Z-scores. Cross-condition comparisons will be the main effect of interest, comparing no drug to remimazolam.
Functional connectivity | Day/Visit 1: during no-drug condition MRI scan, during remimazolam MRI scan
  Whole-brain functional connectivity will be determined in each condition (no-drug and remimazolam). This generates a matrix of cross-correlation values. Cross-condition comparisons will be the main effect of interest, comparing no drug to remimazolam.

CONTACTS AND LOCATIONS:
Overall Officials: Keith M Vogt, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data to share:
  * age, height, weight, sex
  * pain intensity & unpleasantness, ratings
  * observer assessment of sedation at the targeted drug dose
  * Behavioral performance data for long-term memory
  * structural and functional MRI images
Supporting Information: Study Protocol, ICF
Time Frame: After analysis is complete and results have been published, all the above data will be shared in de-identified format, linked together by an assigned subject number.
Access Criteria: Data will be shared via a publicly-accessible online platform that allows user download at no cost.